CLINICAL TRIAL: NCT06431893
Title: An Open-Label, Phase 3 Long-Term Extension (LTE) Study To Assess The Safety, Tolerability, And Efficacy Of Treatment With Pegtibatinase In Participants With Classical Homocystinuria (HCU) Due To Cystathionine Beta Synthase Deficiency (ENSEMBLE)
Brief Title: A Phase 3 Long-term Extension Study to Assess the Long-term Safety and Efficacy of Pegtibatinase Treatment in Participants ≥5 to ≤65 Years of Age With Classical Homocystinuria (HCU) (ENSEMBLE)
Acronym: ENSEMBLE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVTX-TVT058-302
Record Dates: First submitted 2024-05-08; First posted 2024-05-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Homocystinuria
Keywords: Classical homocystinuria; HCU; Cystathionine Beta Synthase Deficiency
MeSH Terms: conditions — Homocystinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- pegtibatinase (Experimental)
  Interventions: Drug: Pegtibatinase

INTERVENTIONS:
Drug: Pegtibatinase — Full Target Dose of pegtibatinase BIW
  Other Names: OT-58; TVT-058

SUMMARY:
The goal of this long-term extension (LTE) study is to evaluate the safety and efficacy of pegtibatinase in patients with classical homocystinuria (HCU). Patients who are active in the Phase 1/2 COMPOSE study or those who complete the 24 weeks of treatment in the Phase 3 HARMONY are eligible to participate.

Participants will be in this clinical study for up to about 13 months including:

* a treatment period of up to 104 weeks
* a 4-week safety follow-up period

DETAILED DESCRIPTION:
Overall Design:

This is a global, multicenter, single-arm, open-label study. Participants who meet all eligibility criteria may transition from other pegtibatinase studies and enroll into this LTE study for long-term safety, efficacy, and clinical assessments of pegtibatinase treatment.

All participants will follow a protocol of self-administration of pegtibatinase unless exempted. During the ENSEMBLE study, an optional protein tolerance modification (PTM) sub-study will also be conducted for eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants active in the COMPOSE study or who completed the 24-week blinded period on the full target dose of study intervention in the Phase 3 HARMONY study

Exclusion Criteria:

* Participant permanently discontinued from study intervention treatment in a previous pegtibatinase study due to serious AE (SAE) or intolerance

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent AEs | Week 1 - Week 108
  Incidence of treatment-emergent AEs
Hypermethioninemia | Week 1 - Week 108
  Incidence of hypermethioninemia
Hypomethioninemia | Week 1 - Week 108
  Incidence of hypomethioninemia
Dietary Protein Rescue | Week 1 - Week 108
  Proportion of participants requiring dietary protein rescue for participants with hypomethioninemia

SECONDARY OUTCOMES:
Total Homocysteine (tHcy) Levels | Week 1 - Week 108
  Relative and absolute changes from baseline in tHcy levels

CONTACTS AND LOCATIONS:
Overall Officials: Michael Imperiale, MD, Study Director — Travere Therapeutics, Inc.
Locations (4):
- United States (4):
  - Travere Investigational Site, Portland, Maine
  - Travere Investigational Site, New York, New York
  - Travere Investigational Site - Virtual Site, Morrisville, North Carolina
  - Travere Investigational Site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to datarequest@travere.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Travere reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication.
Access Criteria: Requires submission and approval of intended use and a data sharing agreement.